CLINICAL TRIAL: NCT04028206
Title: Elastic-band Resistance Exercise or Vibration Treatment With Hydroxymethylbutyrate (HMB) Supplement for Sarcopenic Older People
Brief Title: Resistance Exercise or Vibration With HMB for Sarcopenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof CHOW Kwoon-ho, Simon, Research Assistant Professor of Orthopaedics and Traumatology, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CREC 2018.602
Record Dates: First submitted 2019-07-18; First posted 2019-07-22 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Sarcopenia
Keywords: vibration treatment; sarcopenia; elastic-band resistance; hydroxymethylbutyrate; elderly; randomized control trial
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): No intervention on sarcopenic subjects screened (based on the AWGS definition).
- Exercise + HMB Group (Active Comparator): Sarcopenic subjects on combined treatment of elastic-band exercise and HMB supplementation
  Interventions: Dietary Supplement: Hydroxymethylbutyrate; Behavioral: Elastic-band Exercise
- Vibration Treatment + HMB Group (Active Comparator): Sarcopenic subjects on combined treatment of vibration treatment and HMB supplementation
  Interventions: Dietary Supplement: Hydroxymethylbutyrate; Device: Low-magnitude High Frequency Vibration (LMHFV)

INTERVENTIONS:
Dietary Supplement: Hydroxymethylbutyrate — Hydroxymethylbutyrate supplementation at 3.0 g/day with dietary advice.
  Arms: Exercise + HMB Group; Vibration Treatment + HMB Group
Device: Low-magnitude High Frequency Vibration (LMHFV) — Low-magnitude High Frequency Vibration is a non-invasive biophysical intervention which provides mechanical stimulation with no reported adverse effects. Our previous studies on bone showed that LMHFV can help boost the patients' bone mineral density (BMD) and muscle health.
  Other Names: Vibration treatment
  Arms: Vibration Treatment + HMB Group
Behavioral: Elastic-band Exercise — Subjects enrolled in the elastic-band exercise group will be instructed with 1 session of group training (at baseline) and 1 follow-up home visit (at 4 weeks) including instructions on 5-10 min warm-up and cool-down routines, 30 min chair-based resistance exercises using Thera-Bands as previously reported with training to both upper and lower body muscle groups including both hand and knee extensor muscles. The subjects will be instructed to perform the instructed exercises 3 times per week, one hour after HMB intake, for 12 weeks. The elastic band strengths will be progressively increased from 1.3 kg to 2.1 kg (yellow to green) of tensional force as instructed by a qualified coach in our project team based on each subject's "multiple repetition maximum", where multiple repetition maximum is defined by reaching fatigue by 8 repetitions of stretching.
  Arms: Exercise + HMB Group

SUMMARY:
Sarcopenia is a geriatric syndrome characterised by the progressive loss of skeletal muscle mass and function with a risk of adverse outcomes. In Hong Kong, the prevalence of sarcopenia in community-dwelling older people was 9%. According to a meta-analysis on the effect of sarcopenia on health outcomes in older people, sarcopenia significantly increased hazard ratios of falling by 3.23×, functional decline by 3.03× and fracture risk by up to 3.75×, thus making sarcopenia a major risk factor for fragility fractures.

Elastic-band exercise alone was shown to enhance skeletal muscle mass, performance and gait speed. Low-magnitude high-frequency vibration (LMHFV) was shown to be effective in enhancing muscle strength, balancing ability and reducing fall risk. HMB supplementation is advantageous due to its simplicity in administration and found to be effective in maintaining total lean mass, appendicular lean mass, leg and arm lean masses.

The objective of this study is to evaluate the effectiveness of elastic-band exercise or vibration treatment in combination with HMB supplementation on the control of sarcopenia by a single-blinded randomized controlled study.

Community-dwelling older people failing the sarcopenia screening according to the Asian Working Group on Sarcopenia (AWGS) will be recruited and randomized to (1) control, (2) Exercise + HMB or (3) LMHFV + HMB group by envelope drawing of computer-generated random numbers. Control group will be given promotional materials of sarcopenia and will not receive any intervention. The Exercise + HMB group will be instructed to take a thirty-minute home-based elastic band exercise practiced for 30 mins per day, 3 times per week for 3 months. The LMHFV + HMB group will be assigned to participating community centres and receive vibration treatment at 35Hz, 0.3g (peak to peak magnitude), displacement of <0.1mm, for 20 min/day, at least 3 days/week for 3 months. Both HMB treatment groups will given 3.0 g/day for 3 months. Outcome assessments will be performed at baseline and end-point of 3 months. Outcome assessor and statistician will be blinded to group allocation.

Muscle strength in the lower extremity will be the primary outcome. Muscle strength in the upper extremity, gait speed, muscle mass (based on AWGS definition), functional performance in terms of balancing ability and time-up-and-go test, quality of life by short-form 36 will be taken as secondary outcomes.

DETAILED DESCRIPTION:
Sarcopenia is a geriatric syndrome characterised by the progressive loss of skeletal muscle mass and function with a risk of adverse outcomes. In Hong Kong, the prevalence of sarcopenia in community-dwelling older people was 9%. According to a meta-analysis on the effect of sarcopenia on health outcomes in older people, sarcopenia significantly increased hazard ratios of falling by 3.23×, functional decline by 3.03× and fracture risk by up to 3.75×, thus making sarcopenia a major risk factor for fragility fracture.

A recent study reported a randomized controlled trial (RCT) of 3-month intervention of elastic-band exercise alone has shown significant enhancement in skeletal muscle mass by a 0.7 kg gain and a better performance demonstrated by 0.14 m/s faster gait speed. This project targets to investigate the application of elastic-band exercise for older people to carry out at home for sarcopenia intervention.

Low-magnitude high-frequency vibration (LMHFV) has previously shown to be effective in enhancing muscle strength, balancing ability and reducing fall risk in a RCT involving 710 subjects. Community-dwelling older people treated at 35 Hz, 0.3 g and 20 minutes per day for 18-months showed reduced hazard ratio for fall or fracture (HR=0.56, 95% CI at 0.40-0.78, p=0.001), 2.46 kg increase in quadriceps strength (95% CI at 1.70-3.22, p<0.001) and overall statistically significant improvements in balancing ability.

HMB supplementation is advantageous due to its simplicity in administration compared to various other schemes. In a RCT on the efficacy of HMB supplementation on 10-day bed-rested older adults aged 60-76, 3.0-g/day was found to be effective in maintaining total lean mass, appendicular lean mass, leg and arm lean masses with significant differences.

The objective of this study is to evaluate the effectiveness of elastic-band exercise or vibration treatment in combination with HMB supplementation on the control of sarcopenia by a single-blinded randomized controlled study.

Community-dwelling older people failing the sarcopenia screening according to the Asian Working Group on Sarcopenia (AWGS) will be recruited and randomized to (1) control, (2) Exercise + HMB or (3) LMHFV + HMB group by envelope drawing of computer-generated random numbers. Control group will be given promotional materials of sarcopenia and will not receive any intervention. The Exercise + HMB group will be instructed to take a thirty minute home-based elastic band exercise practiced for 30 mins per day, 3 times per week for 3 months. The LMHFV + HMB group will be assigned to participating community centres and receive the vibration treatment at 35Hz, 0.3g (peak to peak magnitude), displacement of <0.1mm, for 20 min/day, at least 3 days/week for 3 months. Both HMB treatment groups will given 3.0 g/day for 3 months. Outcome assessments will be performed at baseline and end-point of 3 months. Outcome assessor and statistician will be blinded to group allocation.

Muscle strength in the lower extremity will be the primary outcome. Muscle strength in the upper extremity, gait speed, muscle mass (based on AWGS definition), functional performance in terms of balancing ability and time-up-and-go test, quality of life by short-form 36 will be taken as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 65 years old or above
* failing the sarcopenia screening based on the AWGS definition:

  1. hand-grip strength (male at <26 kg, female at <18kg),
  2. gait speed test (<0.8m/s), and/or height-adjusted skeletal muscle mass by bio-impedance analysis (BIA, male at <7kg/m^2 and female at <5.4kg/m^2) defined by appendicular skeletal muscle mass/height^2.

Exclusion Criteria:

* pathological bone diseases
* chronic inflammatory conditions known to affect muscle metabolism; including diabetes, rheumatoid arthritis
* neurological conditions affecting normal gait
* dependent ambulatory capability
* subjects taking regular guided exercise programmes of more than three times per week
* subjects with cardiovascular concern such as with pace-maker in-situ or malignancy
* chair-bound or bed-bound subjects
* recovering from fractures/surgeries or with implants (affecting DXA scan)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2019-09-04 (Actual); Primary Completion 2023-07-29 (Estimated); Study Completion 2023-07-29 (Estimated)

PRIMARY OUTCOMES:
Muscle strength in the lower extremity | 3 months, change is being assessed.
  Quadriceps muscle strength will be measured at the maximum of the quadriceps muscle contraction by a dynamometer. Participants will be instructed to seat on a chair with the knee and hip flexed at 90 degrees and pelvis fixed. The peak isometric forces will be measured 3 times on each leg and the maximum will be taken.

SECONDARY OUTCOMES:
Balancing ability | 3 months, change is being assessed
  Biodex Balance System SD (BioSway, Biodex Medical Systems, USA) will be used to measure the balancing ability of the subjects. This is a verified assessment tool to measure the angular excursion of subject's center of gravity during movement. Parameters of balancing ability include reaction time, movement velocity, maximum/end-point excursion and directional control in limit of stability test.
Timed-up-go test (TUG) | 3 months, change is being assessed
  Time will be recorded for participants to rise from a chair, walk 3 meters, turn around, and walk back to the chair then sitting down.
Dual energy x-ray absortiometry (DXA) | 3 months, change is being assessed.
  Whole body muscle mass measurement
Gait speed | 3 months, change is being assessed.
  A 6-meter-walk test will be used to calculate the gait speed of the participant.
Muscle strength in the upper extremity | 3 months, change is being assessed.
  Handgrip strength will be measured by a dynamometer (5030JI, JAMAR, USA) on each hand of the subject. Participants will be instructed to hold the device with the arm at right angle and elbow to the side of the body.
Quality of life by short-form-36 | 3 months, change is being assessed.
  Health-related quality of life will be assessed by the validated Chinese version of the 36-item Short-Form Health Survey (SF-36).

CONTACTS AND LOCATIONS:
Locations (1):
- Evangelical Luthera Church Social Service - Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Data may be obtained from a third party and are not publicly available. Individual participant data that underlie the results reported in this article will be made available after deidentification .
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Individual participant data will be made available beginning 3 months and ending 3 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal may access data to achieve aims in the approved proposal. Data requestors should direct their proposals to no-fall@ort.cuhk.edu.hk and data will be available after signing a data access agreement.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Background] Stout JR, Smith-Ryan AE, Fukuda DH, Kendall KL, Moon JR, Hoffman JR, Wilson JM, Oliver JS, Mustad VA. Effect of calcium beta-hydroxy-beta-methylbutyrate (CaHMB) with and without resistance training in men and women 65+yrs: a randomized, double-blind pilot trial. Exp Gerontol. 2013 Nov;48(11):1303-10. doi: 10.1016/j.exger.2013.08.007. Epub 2013 Aug 24. PMID 23981904
- [Background] Leung KS, Li CY, Tse YK, Choy TK, Leung PC, Hung VW, Chan SY, Leung AH, Cheung WH. Effects of 18-month low-magnitude high-frequency vibration on fall rate and fracture risks in 710 community elderly--a cluster-randomized controlled trial. Osteoporos Int. 2014 Jun;25(6):1785-95. doi: 10.1007/s00198-014-2693-6. Epub 2014 Mar 28. PMID 24676848
- [Background] Yu R, Wong M, Leung J, Lee J, Auyeung TW, Woo J. Incidence, reversibility, risk factors and the protective effect of high body mass index against sarcopenia in community-dwelling older Chinese adults. Geriatr Gerontol Int. 2014 Feb;14 Suppl 1:15-28. doi: 10.1111/ggi.12220. PMID 24450557
- [Background] Sayer AA. Sarcopenia. BMJ. 2010 Aug 10;341:c4097. doi: 10.1136/bmj.c4097. No abstract available. PMID 20699307
- [Background] Beaudart C, Zaaria M, Pasleau F, Reginster JY, Bruyere O. Health Outcomes of Sarcopenia: A Systematic Review and Meta-Analysis. PLoS One. 2017 Jan 17;12(1):e0169548. doi: 10.1371/journal.pone.0169548. eCollection 2017. PMID 28095426
- [Background] Chen LK, Liu LK, Woo J, Assantachai P, Auyeung TW, Bahyah KS, Chou MY, Chen LY, Hsu PS, Krairit O, Lee JS, Lee WJ, Lee Y, Liang CK, Limpawattana P, Lin CS, Peng LN, Satake S, Suzuki T, Won CW, Wu CH, Wu SN, Zhang T, Zeng P, Akishita M, Arai H. Sarcopenia in Asia: consensus report of the Asian Working Group for Sarcopenia. J Am Med Dir Assoc. 2014 Feb;15(2):95-101. doi: 10.1016/j.jamda.2013.11.025. PMID 24461239
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Zhu LY, Chan R, Kwok T, Cheng KC, Ha A, Woo J. Effects of exercise and nutrition supplementation in community-dwelling older Chinese people with sarcopenia: a randomized controlled trial. Age Ageing. 2019 Mar 1;48(2):220-228. doi: 10.1093/ageing/afy179. PMID 30462162
- [Background] Deutz NE, Pereira SL, Hays NP, Oliver JS, Edens NK, Evans CM, Wolfe RR. Effect of beta-hydroxy-beta-methylbutyrate (HMB) on lean body mass during 10 days of bed rest in older adults. Clin Nutr. 2013 Oct;32(5):704-12. doi: 10.1016/j.clnu.2013.02.011. Epub 2013 Mar 4. PMID 23514626
- [Derived] Chow SK, Chim YN, Cheng KY, Ho CY, Ho WT, Cheng KC, Wong RM, Cheung WH. Elastic-band resistance exercise or vibration treatment in combination with hydroxymethylbutyrate (HMB) supplement for management of sarcopenia in older people: a study protocol for a single-blinded randomised controlled trial in Hong Kong. BMJ Open. 2020 Jun 30;10(6):e034921. doi: 10.1136/bmjopen-2019-034921. PMID 32606057
- See also: 2016 Population By-census. Thematic Report: Older Persons. Hong Kong.: Census and Statistics Department; 2018. — https://www.censtatd.gov.hk/hkstat/sub/sp459.jsp?productCode=B1120105